CLINICAL TRIAL: NCT06851962
Title: Single-blinded, Double-arm, Controlled, Randomized, Multicentre Clinical Trial to Evaluate the Impact of Pharmacogenetic-guided Treatment in Patients With Insufficiently Controlled Type 2 Diabetes
Brief Title: Impact of Pharmacogenetic-Guided Treatment on Type 2 Diabetes Clinical Trial
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EPHIC-DIA2; 2025-520686-46-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-30; First posted 2025-02-28 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Pharmacogenetics; Diabetes type 2; uncontrolled diabetes; hyperglycemia; hypoglycemia; dyslipemia; personalized medicine; genomics; Precision Medicine
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Hypoglycemia | interventions — Metformin; dulaglutide; semaglutide; empagliflozin; Canagliflozin; dapagliflozin; Pioglitazone; Sitagliptin Phosphate; Vildagliptin; Linagliptin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pharmacogenetic-guided treatment (Experimental): Patient treatment will be selected according to previously identified genetic variations. Study treatments and posology from enrollment to the end of treatment at Week 24 can be:
  1. Metformin (daily dose 2000 mg).
  2. GLP1 receptor analogs: dulaglutide and semaglutide.
  3. SGLT2 inhibitors: empagliflozin, canagliflozin and dapagliflozin.
  4. Pioglitazone.
  5. DPP4 inhibitors: sitagliptin, vildagliptin and linagliptin. Or a combination of these drugs. Except of metformin, which 2000 mg is the daily dose stablished in this study, for the rest of treatment options, SmPCs guidelines of each treatment will be followed to stablished the daily dose.
  Interventions: Drug: Metformin; Drug: Dulaglutide; Drug: Semaglutide 1.0 mg; Drug: Empagliflozin (BI 10773); Drug: Canagliflozin; Drug: Dapagliflozin; Drug: pioglitazone; Drug: Sitagliptin; Drug: Vildagliptin (Galvus); Drug: linagliptin
- Standard treatment (Active Comparator): Patient treatment will be selected according to clinical guidelines. Study treatments and posology from enrollment to the end of treatment at Week 24 can be:
  1. Metformin (daily dose 2000 mg).
  2. GLP1 receptor analogs: dulaglutide and semaglutide.
  3. SGLT2 inhibitors: empagliflozin, canagliflozin and dapagliflozin.
  4. Pioglitazone.
  5. DPP4 inhibitors: sitagliptin, vildagliptin and linagliptin. Or a combination of these drugs. Except of metformin, which 2000 mg is the daily dose stablished in this study, for the rest of treatment options, SmPCs guidelines of each treatment will be followed to stablished the daily dose.
  Interventions: Drug: Metformin; Drug: Dulaglutide; Drug: Semaglutide 1.0 mg; Drug: Empagliflozin (BI 10773); Drug: Canagliflozin; Drug: Dapagliflozin; Drug: pioglitazone; Drug: Sitagliptin; Drug: Vildagliptin (Galvus); Drug: linagliptin

INTERVENTIONS:
Drug: Metformin — Metformin maximum daily dose 2000 mg
Drug: Dulaglutide — Dulaglutide
Drug: Semaglutide 1.0 mg — Semaglutide
Drug: Empagliflozin (BI 10773) — Empagliflozin
Drug: Canagliflozin — Canagliflozin
Drug: Dapagliflozin — Dapagliflozin
Drug: pioglitazone — Pioglitazone
Drug: Sitagliptin — Sitagliptin
Drug: Vildagliptin (Galvus) — vildagliptin
Drug: linagliptin — linagliptin

SUMMARY:
The goal of this clinical trial is to assess the efficacy of a pharmacogenetics-guided treatment, compared to standard optimized treatment, in patients with inadequately controlled type 2 diabetes. The main questions it aims to answer are:

* Is the disease better controlled when the treatment prescribed is based on the participant's pharmacogenetic profile?
* What medical problems do participants experience while taking the treatment?

Participants will:

* Take the treatment described according to the Summary of Product Characteristics (SmPC).
* Visit the clinic once every 12 weeks for checkups and tests.
* Keep a diary of their symptoms to inform the Investigator.

DETAILED DESCRIPTION:
Rationale:

Type 2 diabetes (T2D) is a growing disease that causes serious complications and represents a significant public health burden. Despite current therapies, many patients fail to achieve adequate glycemic control, highlighting the need for more personalized approaches. This study seeks to demonstrate that pharmacogenetics, which tailors treatments according to patients' genetic variations, can improve disease control, reduce adverse effects, and ultimately optimize healthcare resources, improving patients' quality of life.

Study Design:

This is a Phase IV, multicenter, randomized, controlled, two-arm, crossover clinical trial. The study will include at least 504 patients, who will be randomized in a 1:1 ratio to receive pharmacogenetics-guided treatment or standard treatment for type 2 diabetes. Once proven to meet eligibility criteria, patients will be assigned to a treatment arm and will participate in the study for the next 24 weeks.

Primary Objective:

To evaluate the efficacy of pharmacogenetics-guided treatment, compared to optimized standard treatment, in patients with inadequately controlled type 2 diabetes.

Secondary Objective:

To evaluate pharmacogenetic markers with the effect of treatment administered prior to randomization.

Exploratory Objectives:

* To evaluate the percentage of patients achieving the target of dyslipidemia and its relationship with the genetic variations present in these subjects.
* To evaluate the percentage of patients reaching the blood pressure target and its relationship with the genetic variations present in these subjects.
* To evaluate the incidence and relationship of adverse events of glucose control drugs with genetic variations.

Safety Objective:

To evaluate the safety and tolerability of the glucose control drugs prescribed in each group of patients.

Target Population:

Patients between 40 and 70 years old, with a body mass index (BMI) between 25 and 40 kg/m² and with a diagnosis of type 2 diabetes inadequately controlled (HbA1c between 7% and 9.5%) and receiving standard non-insulin treatment for at least 6 months will be included. Patients will be visited at 12 and 24 weeks from the start of the study.

Statistical Methods:

The sample size was calculated with an alpha risk of 0.05 and a beta risk of 0.1, using a bilateral test. A total of 252 subjects in each group (standard and pharmacogenetics-guided treatment) are required to detect a significant difference in the proportion of patients achieving HbA1c ≤7%. A dropout rate of 10% is expected. Follow-up of patients will be 24 weeks, sufficient time to observe improvements in glycemic control. The goal is to achieve an HbA1c ≤7%, as recommended by the American Diabetes Association. It is estimated that 50% of patients will achieve the target with antidiabetic treatment, and it is assumed that pharmacogenetics-guided treatment will have at least a 15% greater response than conventional treatment, due to genetic variations.

The main objective is to evaluate the impact of pharmacogenetics-guided treatment in patients with type 2 diabetes, comparing proportions between groups. Analyses will be performed according to the type of variable: Student's t-test or Mann-Whitney for quantitative variables and Fisher's exact test or chi-square tests for qualitative variables. The software used will be R (version 3.6.1), with two-way tests and an alpha risk of 0.05, verifying normality with the Shapiro-Wilk test.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-70 years old, included.
2. Body Mass Index (BMI) between 25-40 kg/m².
3. Diagnosis of Type 2 Diabetes (T2D) according to the American Diabetes Association (ADA) criteria.
4. Patients with T2D insufficiently controlled (Hemoglobin A1c (HbA1c) 7-9.5%) with current (≥6 months) "standard of care" treatment, excluding the use of insulin.
5. The subject has provided written informed consent prior to any study-specific procedure.
6. Able and willing to comply with requested study visits and procedures.
7. Contraceptive measures, only for female participants:

   * A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies:
   * Is a woman of non-childbearing potential (WONCBP) OR
   * Is a woman of childbearing potential (WOCBP) and agrees to use a contraceptive method that is highly effective, with a failure rate of <1%, during the study intervention period (to be effective before starting the intervention).

A WOCBP must have a negative urine pregnancy test before the first administration of study intervention.

Exclusion Criteria:

1. Treatment with insulin at the time of screening.
2. HbA1c >9.5% at screening.
3. Treatment with more than 3 glucose-lowering drugs at the time of screening.
4. Chronic renal disease defined as estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m² (many glucose-lowering drugs are not approved or require dosage adjustments for use in these patients) at the screening visit.
5. Hepatic insufficiency, which contraindicates the use of glucose-lowering drugs.
6. Currently receiving treatment in another investigational drug study, or less than 30 days since ending treatment in another investigational drug study.
7. Pregnancy or lactation.
8. Women of childbearing potential with no effective contraceptive methods.
9. New York Heart Association (NYHA) Class III or IV congestive heart failure.
10. Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the subject and investigator's knowledge.
11. Subject is study staff directly involved with the study or is a family member of the investigational study staff.
12. Life expectancy predicted to be <2 years.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of HbA1c ≤7% goal at Week 24 between Pharmacogenetic-Guided and Standard Treatment in Type 2 Diabetes | From baseline to the end of treatment at 24 weeks
  The primary objective is to compare the proportion of patients achieving HbA1c ≤7% at Week 24 between pharmacogenetic-guided treatment arm and standard treatment arm in subjects with insufficiently controlled type 2 diabetes. The null hypothesis is that the proportion of patients achieving this goal is equal in both the pharmacogenetic-guided and standard treatment groups.

SECONDARY OUTCOMES:
Comparison of Pharmacogenetic Markers and Treatment Response Pre-Randomization | Before randomization to the end of treatment at 24 weeks
  Comparison of pharmacogenetic markers with the effect of pre-randomization treatment. This will be measured by analyzing the pharmacogenetic markers before randomization and their relationship to the treatment response. The endpoint will be the comparison between the proportion of patients who achieved HbA1c ≤7% at baseline (excluded from randomization) and those who did not (included for randomization).

OTHER OUTCOMES:
Exploratory Objective (1): percentage of patients achieving the dyslipidemia goal (LDL colesterol/LDL-C <70 mg/dL or <55 mg/Dl) in patients with or without cardiovascular disease (CVD) | From baseline to the end of treatment at 24 weeks
  Percentage of patients achieving the dyslipidemia goal at Week 24, defined as:
  * LDL-C <70 mg/dL in patients without documented CVD at baseline.
  * LDL-C <55 mg/dL in patients with documented CVD at baseline.
  Additionally, the relationship between these outcomes and genetic variations in the subjects will be measured.
Exploratory Objective (3): percentage of patients achieving the goal of <140/90 mmHg systolic and diastolic pressure | From baseline to the end of treatment at 24 weeks
  To evaluate the percentage of patients achieving the goal of blood pressure as defined in the study (<140/90 mmHg at Week 24) and its relationship with genetic variations present in those subjects.
Exploratory Objective (4): glucose-lowering drugs' adverse events | From baseline to the end of treatment at 24 weeks
  To evaluate incidence and relatedness of glucose-lowering drugs' adverse events with genetic variations.
Safety Objective (1): Incidence of Treatment-Emergent Adverse Events (AEs) | From baseline to the end of treatment at 24 weeks
  To evaluate the percentage of patients who experienced treatment-emergent adverse events (AEs) from baseline to Week 24 in each treatment group. This will be measured by comparing the proportion of patients who present AEs related to glucose-lowering drugs between baseline and Week 24.
Safety Objective (2): Incidence of Serious Adverse Events (SAEs) | From baseline to the end of treatment at 24 weeks
  To evaluate the percentage of patients who experienced serious adverse events (SAEs) from baseline to Week 24 in each treatment group. This will be measured by comparing the proportion of patients who present SAEs related to glucose-lowering drugs between baseline and Week 24.
Safety Objective (1): Changes in hepatic function | From baseline to the end of treatment at 24 weeks
  Hepatic function will be assessed by measuring liver enzymes such as GOT, GPT, GGT in U/L.
Safety Objective (2): Changes in renal function (eGFR) | From baseline to the end of treatment at 24 weeks
  Renal function will be assessed by measuring the glomerular filtration rate (eGFR) in mL/min/m².
Safety Objective (3): Changes in renal function (creatinine) | From baseline to the end of treatment at 24 weeks
  Renal function will be assessed by measuring the levels of creatinine (mg/dl).
Safety Objective (4): Changes in biochemistry parameters (glucose) | From baseline to the end of treatment at 24 weeks
  This will be assessed by measuring several biochemistry parameters such as glucose (mg/dl).
Safety Objective (5): Changes in biochemistry parameters (insulin) | From baseline to the end of treatment at 24 weeks
  This will be assessed by measuring several biochemistry parameters such as insulin (mU/L).
Safety Objective (6): Changes in biochemistry parameters (lipid panel) | From baseline to the end of treatment at 24 weeks
  This will be assessed by measuring several biochemistry parameters such as HDL, LDL and total colesterol in mg/l.
Safety Objective (7): Changes in heart rate | From baseline to the end of treatment at 24 weeks
  This will be measured by comparing the heart rate (bpm) from baseline to Week 24 for each treatment group.
Safety Objective (8): Changes in blood pressure | From baseline to the end of treatment at 24 weeks
  This will be measured by comparing the blood pressure (mmHg) from baseline to Week 24 for each treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Martínez Hervás, Doctor, Principal Investigator — Hospital Clínico Universitario de Valencia
Locations (4):
- Spain (4):
  - Hospital Universitario Regional de Málaga, Málaga
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia (HGUV), Valencia
  - Hospital Universitario Rio Hortega de Valladolid (HURH), Valladolid